CLINICAL TRIAL: NCT03743662
Title: A Phase II Trial of the PD-1 Antibody Nivolumab in Combination With Hypofractionated Re-irradiation and Bevacizumab for Recurrent MGMT Methylated Glioblastoma
Brief Title: Nivolumab With Radiation Therapy and Bevacizumab for Recurrent MGMT Methylated Glioblastoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-400
Record Dates: First submitted 2018-11-13; First posted 2018-11-16 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma
Keywords: WHO grade IV; IDH wildtype; MGMT hypermethylation; 18-400; nivolumab; recurrent glioblastoma; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Glioblastoma | interventions — Re-Irradiation; Bevacizumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Recurrent Glioblastoma, No Surgery (Experimental): One cohort is for patients with recurrent GBM who are not undergoing surgical debulking as part of their treatment plan
  Interventions: Radiation: Re-irradiation (RT); Drug: Bevacizumab; Drug: Nivolumab
- Recurrent Glioblastoma, Surgery (Experimental): The second cohort is for patients with recurrent GBM who are undergoing surgery as part of their treatment.
  Interventions: Radiation: Re-irradiation (RT); Drug: Bevacizumab; Drug: Nivolumab; Procedure: Re-resection

INTERVENTIONS:
Radiation: Re-irradiation (RT) — Re-RT will start on day 28 +/- 5 days for 5 fractions of 600cGy every other day over a 2-week period.
Drug: Bevacizumab — Bevacizumab if deemed beneficial by the investigator, will be started at the initiation of re-RT and continued for three doses in the medical arm. Patients in the surgical arm will omit the first bevacizumab dose to assure adequate wound healing after surgery and receive two doses. Bevacizumab will be dosed at 10mg/kg and given intravenously on day 28 (medical arm only), day 42 and day 56. Following day 56, further bevacizumab doses can be given every two weeks at the discretion of the treating physician.
Drug: Nivolumab — Nivolumab will be started at enrollment and each patient will receive two doses of nivolumab prior to radiation.
  Nivolumab will be dosed at 3mg/kg given intravenously before re-RT (day 1 +/- 5 and 14 +/- 5) and when given with bevacizumab if deemed beneficial by the investigator, (day 28 +/- 5 (medical arm only), day 42 +/- 5, and day 56 +/-5). Nivolumab will be dosed based on body weight while combined with re-radiation and bevacizumab for safety considerations to reduce adverse events. Single agent nivolumab will be given at 240mg flat dose every 2 weeks thereafter until disease progression, withdrawal, adverse event, or death.
Procedure: Re-resection — Re-resection will be performed in the surgical arm at day 14 (+/- 5 days).
  Arms: Recurrent Glioblastoma, Surgery

SUMMARY:
This study is being done to see if adding nivolumab to radiation therapy and bevacizumab can increase the effectiveness of the treatment for recurrent glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmed glioblastoma (WHO grade IV), IDH wildtype confirmed by DNA sequencing
* MGMT hypermethylation in archival tumor biopsy, determined by any CLIAapproved, DNA-based assay
* Prior maximal feasible surgical resection of biopsy
* Prior treatment with radiation and temozolomide chemotherapy
* Pathologic and/or Radiographic evidence of recurrent disease
* Circumscribed enhancing tumor ≤ 5.0 cm in largest diameter (T1 post contrast)
* 1 prior course of radiation therapy
* Age ≥ 18 years
* Karnofsky performance status ≥ 70% or ECOG 0 or 1
* Adequate bone marrow function

  * Hemoglobin ≥ 10g/dL
  * Absolute neutrophil count ≥ 1,500/mm 3
  * Absolute lymphocyte count ≥ 200/mm 3
  * Platelet count ≥ 100,000/mm3
* Adequate liver function

  * Bilirubin <1.5 times upper limit normal (ULN)
  * AST and ALT ≤ 3 times ULN
  * Alkaline phosphatase ≤ 2 times ULN
* Adequate renal function

  * BUN and Creatinine <1.5 times ULN

Exclusion Criteria:

* Infratentorial location of the recurrence
* IDH mutated glioblastoma
* More than one prior tumor recurrence after standard first-line therapy
* Prior radiation to the brain within ≤ 4 months
* Circumscribed enhancing tumor >5.0 cm in largest diameter (T1 post contrast)
* Pulmonary embolus or deep vein thrombosis within preceding 2 months
* Grade 2 or greater congestive heart failure
* Unstable angina, myocardial infarction within past 12 months
* Peptic ulcer, abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within past 6 months
* Nonhealing wound, ulcer or bone fracture
* Prior spontaneous CNS hemorrhage (as determined from clinical history, CT, or MRI)
* Uncontrollable hypertension
* Requiring escalating or chronic supraphysiologic doses of corticosteroids (> 4 mg dexamethasone daily) for control of disease at the time of registration
* Previous or current treatment with an anti-CTLA-4, anti-PD-1, anti-PD-L1, or anti-PDL2 agent.
* Previous or current treatment with bevacizumab
* Hypersensitivity to nivolumab or bevacizumab or any of its excipients
* Diagnosis of immunodeficiency, including Human Immunodeficiency Virus (HIV) or acquired immunodeficiency syndrome (AIDS)
* Known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Known history of active TB (Bacillus Tuberculosis)
* Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Known history of, or any evidence of active, non-infectious pneumonitis.
* Active infection requiring systemic therapy.
* Pregnancy or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Unable to undergo MRI of the brain (i.e. pacemaker or any other contraindication for MRIs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 years
  in participants with recurrent glioblastoma (first recurrence)treated with re-irradiation with concurrent nivolumab (as well as bevacizumab if the investigator feels that the patient benefits from the addition) followed by adjuvant nivolumab in two parallel cohorts.

SECONDARY OUTCOMES:
6 month progression-free survival | 6 months
Median progression-free survival | 2 years
Objective response rate | 2 years
  ORR using the iRANO criteria

CONTACTS AND LOCATIONS:
Overall Officials: Christian Grommes, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (11):
- United States (11):
  - Hartford Healthcare (Data Collection), Hartford, Connecticut
  - Indiana University (Data Collection Only), Indianapolis, Indiana
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Lehigh Valley Health Network (Data Collection Only), Allentown, Pennsylvania
  - University of Vermont Medical Center (Data Collection Only), Burlington, Vermont

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org